CLINICAL TRIAL: NCT05495815
Title: Randomized Clinical Trial Determining Proper Duration of Suppressive Antibiotic Therapy After Total Joint Arthroplasty Debridement, Antibiotics, and Implant Retention
Brief Title: Proper Duration of Suppressive Antibiotic Therapy After Debridement, Antibiotics, and Implant Retention
Acronym: ProperSAT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: OrthoCarolina Research Institute, Inc. (Other); University of Arkansas (Other); OrthoMichigan (Unknown); NYU School of Medicine (Unknown); Sinai Hospital (Unknown); MedStar Health (Other)
Responsible Party: Principal Investigator, Sumon Nandi, Associate Professor, Chief of Adult Reconstruction, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Maryland
Record Dates: First submitted 2022-08-05; First posted 2022-08-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Periprosthetic Joint Infection; Antibiotic Suppression
MeSH Terms: interventions — diamine N-acetyltransferase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 6 months of SAT (Active Comparator): TJA DAIR, followed by 6 weeks of IV antibiotics then 6 months of oral suppressive antibiotic therapy
  Interventions: Drug: 6 months of SAT
- 12 months of SAT (Active Comparator): TJA DAIR, followed by 6 weeks of IV antibiotics then 12 months of oral suppressive antibiotic therapy
  Interventions: Drug: 12 months of SAT
- Indefinite SAT (Active Comparator): TJA DAIR, followed by 6 weeks of IV antibiotics then indefinite oral suppressive antibiotic therapy
  Interventions: Drug: Indefinite SAT

INTERVENTIONS:
Drug: 6 months of SAT — 6 months of oral suppressive antibiotic therapy
  Arms: 6 months of SAT
Drug: 12 months of SAT — 12 months of oral suppressive antibiotic therapy
  Arms: 12 months of SAT
Drug: Indefinite SAT — Indefinite oral suppressive antibiotic therapy
  Arms: Indefinite SAT

SUMMARY:
Multiple studies have demonstrated oral suppressive antibiotic therapy (SAT), after intravenous antibiotics, maximizes reoperation-free survival of total joint arthroplasty (TJA) debridement, antibiotics, and implant retention (DAIR) for acute periprosthetic joint infection (PJI). However, little is known regarding sequelae of SAT after DAIR for PJI. Prior studies have small or heterogeneous patient cohorts, variable antibiotic regimens, arrive at disparate conclusions, and do not establish antibiotic resistance risk.

The investigators propose a prospective randomized controlled multicenter study to expand on findings in a retrospective, multi-center pilot study. Study aims are to evaluate SAT after DAIR of acutely infected primary TJA regarding: 1) adverse drug reactions/intolerance; 2) reoperation for infection; and 3) antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years-old
* underwent DAIR with modular component exchange for acute TJA PJI, as defined by Musculoskeletal Infection Society Criteria, with symptom duration less than 4 weeks
* on postoperative oral SAT for at least 3 months

Exclusion Criteria:

* underwent aseptic revision surgery
* had one-stage, 1.5-stage, or two-stage revision surgery
* did not have postoperative SAT
* did not have follow-up that allowed for evaluation of SAT sequelae

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Reoperation for infection recurrence | 2 years after patient enrollment

SECONDARY OUTCOMES:
Antibiotic resistance, evidenced by change in antimicrobial sensitivity profile, developed by infecting organism after suppressive antibiotic therapy causing infection recurrence | At time of reoperation (within 2 years of patient enrollment)
Adverse drug reaction or intolerance, defined as any symptom or laboratory value derangement requiring a change in, or discontinuation of, antimicrobial therapy | During antibiotic administration (up to 2 years after patient enrollment)
  Antibiotic intolerance is any Grade I sign from CTCAE v5.0, while adverse drug reaction is any Grade 2 sign or higher.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No